CLINICAL TRIAL: NCT00348894
Title: A Phase 2b Long-Term, Randomized, Open-Label, Safety And Tolerability Trial Comparing [S,S]-Reboxetine (PNU-165442g) With Routine Care In Patients With Chronic Painful Diabetic Peripheral Neuropathy (DPN).
Brief Title: [S,S]-Reboxetine Long Term Safety Study In Chronic Painful Diabetic Peripheral Neuropathy.
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: - Study was terminated due to insufficient clinical efficacy observed in previous studies conducted in postherpetic neuralgia.
Sponsor: Pfizer (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer Inc
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: A6061031
Record Dates: First submitted 2006-07-04; First posted 2006-07-06 (Estimated); Last update posted 2011-06-01 (Estimated); Status verified 2011-05

CONDITIONS: Pain
MeSH Terms: conditions — Pain | interventions — O-methyl reboxetine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Open Treatment (Experimental): [S,S]-reboxetine
  Interventions: Drug: [S,S]-Reboxetine
- Standard Care (Other): Standard Care
  Interventions: Drug: Any

INTERVENTIONS:
Drug: [S,S]-Reboxetine — [S,S]-reboxetine
  Arms: Open Treatment
Drug: Any — Any standard of care treatment for DPN
  Arms: Standard Care

SUMMARY:
The purpose of this study is to assess the long-term safety and tolerability of [S,S]-Reboxetine in patients with chronic painful diabetic peripheral neuropathy

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of type 1 or 2 diabetes mellitus, with painful, distal, symmetrical, sensorimotor polyneuropathy
* Patients at screening must have a score >/=40 mm on the pain visual analogue scale

Exclusion Criteria:

* Patients with significant hepatic impairment
* Patients with other severe pain, that may impair the self-assessment of the pain due to DPN

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 136 (Actual)
Dates: Start 2006-07; Primary Completion 2007-10 (Actual); Study Completion 2007-10 (Actual)

PRIMARY OUTCOMES:
Vital signs | duration of study
Physical examination | duration of study
12-lead ECG | duration of study
Hematology/Biochemistry | duration of study
Adverse events | duration of study

SECONDARY OUTCOMES:
Pain Visual Analogue Scale | duration of study
Neuropathic Pain Symptom Inventory | duration of study
Modified Brief Pain Inventory-Short Form | duration of study
Patient Global Impression of Change | duration of study
SF-12 Health Survey | duration of study
EQ-5D | duration of study
Analgesic Treatment Satisfaction Scale | duration of study
Pain-related Medication Utilization | duration of study

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (81):
- United States (23):
  - Pfizer Investigational Site, Birmingham, Alabama
  - Pfizer Investigational Site, Phoenix, Arizona
  - Pfizer Investigational Site, Scottsdale, Arizona
  - Pfizer Investigational Site, Jonesboro, Arkansas
  - Pfizer Investigational Site, Auburn, California
  - Pfizer Investigational Site, Huntington Beach, California
  - Pfizer Investigational Site, Orangevale, California
  - Pfizer Investigational Site, Naples, Florida
  - Pfizer Investigational Site, Winter Park, Florida
  - Pfizer Investigational Site, Honululu, Hawaii
  - Pfizer Investigational Site, Chicago, Illinois
  - Pfizer Investigational Site, Columbia, Missouri
  - Pfizer Investigational Site, Jefferson City, Missouri
  - Pfizer Investigational Site, St Louis, Missouri
  - Pfizer Investigational Site, Omaha, Nebraska
  - Pfizer Investigational Site, Las Vegas, Nevada
  - Pfizer Investigational Site, Reno, Nevada
  - Pfizer Investigational Site, Nashua, New Hampshire
  - Pfizer Investigational Site, Syracuse, New York
  - Pfizer Investigational Site, Greensboro, North Carolina
  - Pfizer Investigational Site, Dallas, Texas
  - Pfizer Investigational Site, Richmond, Virginia
  - Pfizer Investigational Site, Tacoma, Washington
- Pfizer Investigational Site, Buenos Aires, Argentina
- Canada (5):
  - Pfizer Investigational Site, Winnipeg, Manitoba
  - Pfizer Investigational Site, Ottawa, Ontario
  - Pfizer Investigational Site, Toronto, Ontario
  - Pfizer Investigational Site, Laval, Quebec
  - Pfizer Investigational Site, Montreal, Quebec
- Croatia (2):
  - Pfizer Investigational Site, Osijek
  - Pfizer Investigational Site, Split
- Estonia (4):
  - Pfizer Investigational Site, Pärnu
  - Pfizer Investigational Site, Tallinn
  - Pfizer Investigational Site, Tartu
  - Pfizer Investigational Site, Viljandi Mk.
- Finland (4):
  - Pfizer Investigational Site, Helsinki
  - Pfizer Investigational Site, Oulu
  - Pfizer Investigational Site, Seinäjoki
  - Pfizer Investigational Site, Tampere
- Germany (7):
  - Pfizer Investigational Site, Bad Mergentheim
  - Pfizer Investigational Site, Mainz
  - Pfizer Investigational Site, Meissen
  - Pfizer Investigational Site, Münster
  - Pfizer Investigational Site, St.Ingbert
  - Pfizer Investigational Site, Tann I.d. Rhoen
  - Pfizer Investigational Site, Würzburg
- India (6):
  - Pfizer Investigational Site, Hyderabad, Andhra Pradesh
  - Pfizer Investigational Site, Bangalore, Karnataka
  - Pfizer Investigational Site, Maharashtra, Mumbai
  - Pfizer Investigational Site, Ansārinagar, New Delhi
  - Pfizer Investigational Site, Ludhiana
  - Pfizer Investigational Site, Vellore
- Poland (6):
  - Pfizer Investigational Site, Bytom
  - Pfizer Investigational Site, Lodz
  - Pfizer Investigational Site, Lublin
  - Pfizer Investigational Site, Otwock
  - Pfizer Investigational Site, Wroclaw
  - Pfizer Investigational Site, Łask
- Russia (2):
  - Pfizer Investigational Site, Moscow
  - Pfizer Investigational Site, Saint Petersburg
- South Africa (8):
  - Pfizer Investigational Site, Johannesburg, Gauteng
  - Pfizer Investigational Site, Parktown, Gauteng
  - Pfizer Investigational Site, Durban, KwaZulu-Natal
  - Pfizer Investigational Site, Durban, Overport
  - Pfizer Investigational Site, Durban
  - Pfizer Investigational Site, Houghton, Johannesburg
  - Pfizer Investigational Site, Pretoria
  - Pfizer Investigational Site, Soweto
- Sweden (3):
  - Pfizer Investigational Site, Gothenburg
  - Pfizer Investigational Site, Stockholm
  - Pfizer Investigational Site, Umeå
- Ukraine (5):
  - Pfizer Investigational Site, Dnipropetrovsk
  - Pfizer Investigational Site, Donetsk
  - Pfizer Investigational Site, Kharkiv
  - Pfizer Investigational Site, Kyiv
  - Pfizer Investigational Site, Odesa
- United Kingdom (5):
  - Pfizer Investigational Site, Carshalton, Surrey
  - Pfizer Investigational Site, Bath
  - Pfizer Investigational Site, Dundee
  - Pfizer Investigational Site, London
  - Pfizer Investigational Site, Manchester

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A6061031&StudyName=%5BS%2CS%5D-Reboxetine%20Long%20Term%20Safety%20Study%20In%20Chronic%20Painful%20Diabetic%20Peripheral%20Neuropathy.%0A